CLINICAL TRIAL: NCT05797259
Title: RANKL Antibody (Danosumab) for Acute Charcot Neuro-osteoarthropathy Remission in Chronic Kidney Disease
Brief Title: RANKL Antibody for Acute Charcot Neuro-osteoarthropathy
Acronym: DANCN-CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DANCN 01
Record Dates: First submitted 2023-03-06; First posted 2023-04-04 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Charcot Joint of Foot
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Danosumab (Experimental): Danosumab 60mg subcutaneous once at diagnosis
  Interventions: Drug: Danosumab
- Placebo (Placebo Comparator): Similar Volume, and consistency placebo (Normal Saline) subcutaneous once at diagnosis
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Danosumab — 60 mg subcutaneous Danosumab
  Other Names: Drug Arm
  Arms: Danosumab
Other: Normal Saline — Placebo comparator arm
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study's goal was to determine how denosumab 60 mg, combined with total contact casting and restricted weightbearing status, would affect the treatment of acute CN with CKD.

METHODS Participants in the research were those who visited the outpatient foot clinic at PGIMER, CHD in India. During the study period, 446 persons with CN were identified, 102 of whom met the criteria for the first screening, and 78 of whom were ultimately enrolled in the study.

Aim: To assess the clinico-radiological remission of Acute Charcot-neuroarthropathy in patients of CKD.

DETAILED DESCRIPTION:
Participants attending the outpatient diabetic foot facility of tertiary care hospital in North India were assessed for active CN. An active CN of the foot was considered in the presence of localised erythema, edoema, and a temperature differential of more than 20C compared to a similar location on the opposite foot. Participants were diagnosed with "active on chronic" CN if they met the requirements for active CN in the context of foot deformities suggestive of chronic CN (rocker bottom deformity). Those with self-reported diabetes or those who were already receiving treatment for diabetes, with an estimated glomerular filtration rate (eGFR) <60 ml/min/m2 (CKD-EPI equation) and more than 500 mg of urine protein/24 hours were considered as having diabetic CKD. Patients with active pedal ulcer, inactive charcot foot, peripheral vascular disease (ankle brachial index ABI <0.9), prior exposure to medications affecting bone metabolism particularly bisphosphonates, teriparatide, denosumab or steroids in the past 12 months, hypocalcemia, active malignancy, CKD on dialysis and pregnancy or lactating women were excluded. The study was conducted in accordance with the Declaration of Helsinki and its amendments, the International Conference on Harmonization Good Clinical Practice guidelines, and its applicable regulatory requirements. All participants provided their signed, fully informed consent and study protocol was approved by the institutional Ethics Committee ref INT/IEC/SPE-1664.

The foot temperature was determined by an infrared dermal thermometry [(FLIR Systems Inc, Orlando, USA) with a pixel resolution of 4800 (80*60), thermal sensitivity of 0.15 C, and a detection range of -20 C to 250 C] after 30 minutes of removing footwear or cast. X-ray and/or magnetic resonance imaging (MRI) were used to confirm the diagnosis of an active CN (3T scanner Siemens MagnetromVerio). The involved area of foot was classified anatomically for pattern of involvement using the Sanders-Frykberg classification. Clinical information was documented, including the duration of the symptoms, duration of diabetes, concomitant microvascular and macrovascular complications. Comprehensive neurological testing included vibration perception threshold (VPT>25 mV was considered abnormal) by biothesiometer-Vibrometer-VPT1 (Diabetik Foot Care, Madras Engineering Service, India), perception of 10-g monofilament at 5 standardised plantar locations, and ankle reflex.

Interventions:

Participants were randomly assigned in 1:2 ratio to receive either injection denosumab 60 gm (Group A) or equal volume of normal saline (Group B) subcutaneous over abdomen as a single dose (denosumab and normal saline were provided in similar looking syringe). The investigator administering the treatment, radiologist and the patient were blinded to treatment allocation. A conventional below knee, non-walking, non-removable fibreglass total contact cast (TCC) were provided to all participants irrespective of the group allocation for offloading.

Procedures:

Participants visited the study site initially during screening, randomization and subsequently four weekly for the monitoring of foot temperature. During randomization visit, blood samples were drawn for HbA1c, renal functions, calcium, phosphate and vitamin D. An average of three temperature readings at the afflicted site of the foot were taken and temperature difference (0C) were noted. The study drug or placebo were administered by blinded investigator and TCC was provided. Subsequently, during 4-weekly follow up visits the cast was removed for 30 minutes and skin temperature (mean of three readings) difference was noted. A change of cast was performed four weekly or earlier to avoid "pistoning" effect caused by the edema diminution until clinical remission. Patients with vitamin D deficiency (25 (OH)D3<30 ng/ml were supplemented with weekly oral cholecalciferol 60,000 IU for 8 weeks , then monthly till end of follow up.

A temperature difference of <2C between the afflicted foot and a similar site on the other foot documented twice (four weeks apart) along with the absence of signs of inflammation was considered "clinical remission" of active CN.

Following the clinical remission of active CN, the TCC shall be discontinued, and participants received cast walkers or customised footwear. Subsequently, foot examination shall be performed to monitor for the recurrence of CN (foot temperature assessment), the occurrence of deformities or ulcers (clinical examination), new-onset fractures (radiological assessment)or amputation for a minimum duration of 48 weeks following remission.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Active Charcot neuroarthropathy of either left or right foot
* Chronic Kidney disease defined as eGFR<60 ml/min/m2 and/or Urine protein >300 mg/day
* Presence of all

Exclusion Criteria:

* Active Pedal ulcer
* Active malignancy
* Hypocalcemia
* Primary Hyperparathyroidism
* Pregnancy and Breast Feeding
* Prior treatment with anti-RANKL antibody
* On corticosteroids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Remission of acute charcot | 48 week
  Proportion of patients achieving remission

SECONDARY OUTCOMES:
Remission duration | 48 week
  Remission duration in weeks or months
Recurrence of CN | 48 week
  Recurrence of active CN defined by temperature >2 C in the affected foot after documenting remission
Mortality | Death due to any cause during the study duration
  All cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Deptt of Endocrinology, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No